CLINICAL TRIAL: NCT05647174
Title: Developing a Magnetic-POCUS-assisted Bronchoscopy in Difficult Endotracheal Intubation
Brief Title: MGPOCUS Assisted Bronchoscopy in Difficult Endotracheal Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MGPOCUS-DTI
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGPOCUS-assisted bronchoscope-guided intubation (Active Comparator)
  Interventions: Procedure: MGPOCUS-assisted bronchoscope-guided intubation
- Bronchoscope-guided Intubation (Experimental)
  Interventions: Procedure: Bronchoscope-guided intubation

INTERVENTIONS:
Procedure: MGPOCUS-assisted bronchoscope-guided intubation — Application of ultrasound instruments that can detect magnetic signals to determine the position of the magnetised bronchoscopy to guide the direction of its advancement and thus optimise difficult endotracheal intubation.
  Arms: MGPOCUS-assisted bronchoscope-guided intubation
Procedure: Bronchoscope-guided intubation — Routine bronchoscope- guided intubation.
  Arms: Bronchoscope-guided Intubation

SUMMARY:
Introduction Endoracheal intubation (ETI) is a crucial but risky procedure, especially among patients with suspected difficult endotracheal intubation (DTI). Bronchoscopy, as an improved technique commonly used in DTI, might encounters the difficulties of visualization. The magnetic point-of-care ultrasound (MGPOCUS) not only provide an novel visualization from outside, but also enable the estimation of relative position and trajectory of bronchoscopy. The study aims to evaluate the efficiency of MGPOCUS assisted bronchoscopy in time taken to the first-attempt success, the first-attempt and overall success of ETI, complications and satisfaction of visualization among patients suspected with DTI.

Methods and analysis The current study is a randomized, parallel-group, single-blinded, single-center study. Participants (n=350) will be recruited by primary anesthesiologist and randomized to groups of ETI with bronchoscopy or MGPOCUS assisted bronchoscopy. The primary outcome is time taken to the first-attempt success ETI. Secondary outcomes include procedure time, the first-attempt and overall success, complications and satisfaction of visualization. Cox regression with the Bonferroni correction and the linear mixed regression will be used to analysis the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 85 years old.
* Requiring ETI.
* Anticipated DTI meets one or more positive findings in the airway evaluation, including history, examination, and appropriate investigations of anatomy .
* Signed written informed consent.
* Willingness for the primary anesthesia team to participate.

Exclusion Criteria:

* Anterior neck lesions (masses, lacerations, or subcutaneous emphysema).
* A history of neck operation or tracheotomy.
* Allergies to ultrasound coupling gel.
* At risk of pulmonary or cardiovascular complications during intubation with flexible bronchoscope, including severe hypoxemia, severe pulmonary hypertension, unstable or severe obstructive airway disease.
* At risk of bleeding during bronchoscope, including anticoagulants or coagulopathy, renal insufficiency, and superior vena cava syndrome.
* High risk of aspiration.
* Current pregnancy.
* Patient unable to cooperate (for awake intubation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to success | At once after performing intubation at the first attempt and confirming successful endotracheal intubation by capnography
  Time taken in seconds to successful intubation at the first-attempt

SECONDARY OUTCOMES:
Procedure time | Whiler performing intubation.
  Accumulation of every attempts (no more than 2) from bronchoscope passage of teeth to tube well placed.
The first-attempt success | At once after the first-attempt and confirmed by capnography..
  Intubation at the first attempt is whether successful or failure, confirmed by capnography.
Overall success | At once after procedure and confirmed by capnography.
  Intubation is whether successful or failure within no more than 2 attempts and no more than 600 seconds, confirmed by capnography.
Number of attempts | While performing the procedure
  Number of attempts to fulfill intubation
Satisfaction with visualizaiton | At once after every attempt before confirmed by capnography
  Satisfaction with visualization estimated by performers.
Intubation relative complications | At once after performing procedure and after extubation.
  Including desaturation (<90%), obvious trauma ,bloody secretions, post-extuvation hoarseness and sore throat.

CONTACTS AND LOCATIONS:
Locations (1):
- Peing Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Data is available upon request from the corresponding author after the completion of the study.

REFERENCES:
- [Derived] Tian Y, Fei Y, Bai B, Cui X, Zhang Y, Wang C, Yu C, Huang Y. Developing a magnetic POCUS-guided bronchoscope for patients with suspected difficult endotracheal intubation in a general tertiary hospital: protocol for a randomised controlled study. BMJ Open. 2023 Jun 27;13(6):e071325. doi: 10.1136/bmjopen-2022-071325. PMID 37369409